CLINICAL TRIAL: NCT05674617
Title: PTSD Treatment for Veterans With Serious Mental Illness to Improve Functional Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4272-W; 1IK2RX004272-01A1 (NIH)
Record Dates: First submitted 2022-12-02; First posted 2023-01-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Stress Disorders, Post-Traumatic; Mental Disorders
Keywords: Stress Disorders, Post-Traumatic; Mental Disorders; Culturally responsive assessment
MeSH Terms: conditions — Stress Disorders, Traumatic; Mental Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: randomized controlled trial (RCT)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Written Exposure Therapy (WET) (Experimental): 5 individual therapy sessions of WET via video telehealth
  Interventions: Behavioral: Written Exposure Therapy
- PTSD Education Control (Active Comparator): 5 individual sessions of PTSD psychoeducation via video telehealth
  Interventions: Behavioral: PTSD Education

INTERVENTIONS:
Behavioral: Written Exposure Therapy — WET will be conducted in accordance with the Written Exposure Therapy for PTSD: A Brief Treatment Approach for Mental Health Professionals Manual and the VA evidence-based practice (EBP) rollout training.
  Other Names: WET
  Arms: Written Exposure Therapy (WET)
Behavioral: PTSD Education — The 5-session PTSD psychoeducation and skills protocol we will be utilizing for our PTSD education control condition was developed by PTSD clinical team (PCT) clinicians at the Washington DC VA Medical Center as a group protocol for Veterans admitted to the PCT and who were on the waitlist for individual therapy with an EBP for PTSD. The "PTSD 101" protocol consists of psychoeducation on topics related to PTSD symptoms and an introduction to PTSD-related coping skills. Its duration and structure will be similar to WET (5 weekly individual 50-minute sessions). To parallel the time an attention given in individual WET sessions more closely, participants will quietly review any written materials or videos that are a part of the manualized curriculum for 30 minutes of the session, bookended by a 10-minute check-in with their provider on symptoms and introduction to new materials at the start of session and another 10-minute debrief of reviewed materials at the end of session.
  Arms: PTSD Education Control

SUMMARY:
PTSD is common among Veterans with serious mental illness (SMI). Co-occurring PTSD and SMI lead to poorer mental health and physical functioning than either diagnosis alone. Despite known high prevalence rates of PTSD in SMI populations as well as disparities in prevalence and treatment use for Black, Indigenous, and other people of color (BIPOC), little research has been done to: a) evaluate leading treatments for PTSD in individuals with SMI, and b) develop culturally responsive methods to integrate with PTSD treatments for SMI Veterans. This study aims to address research and clinical gaps by: a) testing the feasibility and acceptability of Written Exposure Therapy (WET), a VA evidence-based psychotherapy for PTSD in Veterans with SMI, and b) incorporating culturally responsive assessment methods. Results from this study will inform whether WET and culturally responsive assessment are feasible to implement, acceptable to Veterans with SMI, and worth examining in standard or optimized form in a larger clinical trial.

DETAILED DESCRIPTION:
Project Background: PTSD is prevalent among Veterans and others with serious mental illness (SMI), contributing to substantial mental and physical health impairments. Written Exposure Therapy (WET) is a new evidence-based practice for PTSD that may have special clinical utility for Veterans with SMI and PTSD. However, such Veterans have been largely excluded from PTSD clinical trials, and no WET trials to date have focused on an SMI population. Further, there are significant race and ethnicity disparities in PTSD and SMI prevalence and treatment, even in Veterans Health Administration. For instance, persistence and chronicity of SMI and PTSD are higher for Black, Indigenous, and other people of color (BIPOC) underlining the need for PTSD EBPs to be delivered in culturally responsive ways.

Project Objectives: The proposed CDA-2 research will address research and clinical gaps by integrating culturally responsive assessment methods and testing the feasibility and acceptability of WET among Veterans with SMI and PTSD. The first step of this research will focus on administering culturally responsive assessments and WET to Veterans with PTSD and SMI in a training trial (n = 10), including qualitative interviews exploring participants' experiences with and views of these instruments and WET. The second step will involve completing a small randomized controlled trial of WET to examine feasibility, acceptability, and fidelity of WET, and to preliminarily explore changes to clinical outcomes and functioning among 48 Veterans randomized to WET (n = 32) vs. a PTSD psychoeducation control intervention (n = 16). We will assess rates of recruitment, initial intervention engagement, and session attendance (feasibility); Veteran satisfaction with WET (acceptability); and preliminarily explore response to WET. The final step of this research will involve conducting a process evaluation to consider ways to optimize WET for future clinical trials to improve functional recovery for Veterans with SMI. This evaluation will synthesize information from: 1) WET interventionist notes and 2) qualitative interviews with a subset of Veterans in the WET condition (n = 15).

Project Methods: This project will include: 1) delivering WET with the CFI during a training trial followed by qualitative interviews with Veterans with PTSD and SMI; 2) completing a randomized control trial (RCT) with 48 Veteran participants, monitoring fidelity, feasibility, and acceptability; and 3) studying Veterans' experiences of WET and culturally responsive assessment methods through qualitative interviews. The investigators will measure functional outcomes during the RCT at baseline, post-treatment and 3-month follow-up using clinician-rated and self-report questionnaires for preliminary exploratory analysis, preparatory to a future full RCT if WET proves promising.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in outpatient mental health services within the VAMHCS (including general outpatient Mental Health Clinic (MHC), Psychosocial Rehabilitation and Recovery Centers (PRRCs), Mental Health Intensive Case Management (MHICM), and PTSD Clinical Teams (PCTs))
* diagnosis of PTSD as confirmed by assessment with the Clinician-administered PTSD Scale for DSM-5 (CAPS-5) past month version
* SMI diagnosis as defined by VHA Directive 1160 (i.e., psychotic spectrum or bipolar disorders) as confirmed by the medical record
* regular telephone access

Exclusion Criteria:

* are engaging in moderate-to-severe substance use that would impact their ability to participate and/or would require a higher level of care
* already engaged in trauma-focused EBP for PTSD (e.g., WET, CPT, PE, or EMDR) or completed an EBP for PTSD within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants eligible divided by Individuals approached for recruitment | Through study completion, an average of 1 year
  As a measure of feasibility, the investigators will evaluate recruitment and suitability of eligibility criteria by calculating number eligible participants (e.g., those that passed screening) divided by number potential participants that were approached for recruitment.
Client Satisfaction Questionnaire (CSQ-8) | Post-treatment (~7 weeks)
  Acceptability Full measure title: Client Satisfaction Questionnaire (CSQ-8) Minimum score: 8 Maximum score: 32 Score interpretation: Greater scores indicate greater client satisfaction. Citation: Attkisson, C. C., & Greenfield, T. K. (1994). Client Satisfaction Questionnaire-8 and Service Satisfaction Scale-30. In M. E. Maruish (Ed.), The use of psychological testing for treatment planning and outcome assessment (p. 402-420). Hillsdale, NJ, US: Lawrence Erlbaum Associates, Inc.
Retention and adherence rates | at study completion, approximately 4 years
  As a measure of feasibility, the investigators will calculate percent of randomized who attend first 2 sessions.
Mean number of sessions attended | at study completion, approximately 4 years
  A measure of feasibility via adherence.
Treatment dropout percentage | at study completion, approximately 4 years
  As a measure of feasibility, the investigators will calculate treatment dropout percentage based on the number who dropped out prior to completing treatment divided by the number who engaged.

SECONDARY OUTCOMES:
Clinician-administered PTSD Scale for DSM-5 (CAPS-5) - Past Month Version | Baseline, Post-treatment (~7 weeks), 3-month Follow-up (~19 weeks)
  PTSD symptom improvement Full measure title: Clinician-administered PTSD Scale for DSM-5 (CAPS-5) - Past Month Version Minimum score: 0 Maximum score: 80 Score interpretation: Greater scores indicate greater severity of PTSD symptoms.
  Citation: Weathers, F. W., Blake, D. D., Schnurr, P. P., et al. (2013). The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). Available online from the National Center for PTSD.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline, Post-treatment (~7 weeks), 3-month Follow-up (~19 weeks)
  Health-related functioning Full measure title: World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) Minimum score: 0 Maximum score: 100 Score interpretation: Greater scores indicate greater disability and/or functional impairments.
  Citation: Ustun, T., Chatterji, S., Kostanjsek, N., et al. (2010). Developing the World Health Organization Disability Assessment Schedule 2.0. Bulletin of the World Health Organization, 88(11), 815-823.

CONTACTS AND LOCATIONS:
Overall Officials: Mary K Howell, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No